CLINICAL TRIAL: NCT00385151
Title: The Mechanism of Ischemic Post Conditioning in Humans, Minimizing Reperfusion Injury.
Brief Title: To Compare the Ischemic Pre-conditioning and Post-conditioning on Reperfusion Injury in Humans.
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Principal Investigator, Emory University
Other Study IDs: 0920-2004
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Endothelial Dysfunction
Keywords: Post conditioning

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Reperfusion Injury occurs by the sudden blood flow to the injured and ischemic myocardium during restoration of blood flow either by Mechanical revascularization or thrombolysis. A phenomenon known as Pre-conditioning has been identified to limit the the extent and severity of reperfusion injury but it is very difficult to apply it in patient care setting as timing of acute cardiac or neurologic ischemic event is difficult to reliably predict.

Postconditioning or ischemic postconditioning is well known to attenuate the reperfusion injury. There is enough data that shows the benefit of post conditioning in reducing the reperfusion injury in animals. However postconditioning in humans has not been investigated.

We hypothesize that Post conditioning will attenuate the reperfusion injury and will be comparable to the effect of preconditioning in humans.

DETAILED DESCRIPTION:
Myocardial ischemia is one on the leading causes of mortality and morbidity in the United States. The initial injury to the myocardium is due to a state of imbalance when oxygen demand exceeds supply. This is most pronounced in the cases of sudden total occlusion of a coronary artery that results in myocardial injury and necrosis (AMI). The main stay of the therapy in these cases is the restoration of the flow to the ischemic myocardium by means of reperfusion therapy such as thrombolysis or mechanical revascularization. Interestingly, there is data to suggest that sudden restoration of blood flow to the ischemic myocardium may cause another form of myocardial injury ,known as reperfusion injury.

Although initially controversial, reperfusion injury is now recognized as a distinct entity. This refers to the sudden and brisk reperfusion of ischemic myocardium that may induce injury that was not originally present-paradoxically exaggerating the end result of an ischemic event. Reperfusion injury may increase infarct size, decrease myocardial contractile function and induce or exaggerate vascular endothelial dysfunction. The pathophysiology is not well understood, but some of the effects of reperfusion injury have been attributed to the generation of free oxygen radical and increased oxidative stress possibly related to the abnormalities of the nitric oxide synthase (NOS) enzyme and its byproducts. These cellular events lead to the endothelial dysfunction, a pivotal event in the development of reperfusion injury.

A concept known as pre-conditioning has been identified as a phenomenon that limits the extent and severity of reperfusion injury. Classically, preconditioning refers to the occurrence whereby repeated brief episodes of ischemia preceding a prolonged period of ischemia results in marked diminution of ischemic injury and injury occurring during reperfusion. The mechanism of this ischemic tolerance was thought to be secondary to the recruitment of collateral circulation, as it was noted to develop in patients undergoing serial balloon inflations during angioplasty. The cellular mechanism involved in ischemic preconditioning are not completely understood, but may be related to the attenuation of reperfusion injury. These findings are also corroborated by Kharbanda's group in their findings made after inducing forearm ischemia in 31 healthy volunteers. In an attempt to test the effects of ischemic preconditioning on the attenuation of ischemia-reperfusion injury as it pertains to endothelial function and circulating blood cell function, the forearms of these volunteers were made ischemic for a 20 minutes period using a pneumatic blood pressure cuff to 200 mmHg. This method was then compared to the use of ischemic preconditioning prior to the prolonged 20 minutes ischemic episode. Ischemic preconditioning was induced by inflating the pneumatic cuff to 200 mmhg for 5 minutes and then deflating the cuff. This was repeated for a total of 3 times. Radial artery reactivity testing and blood samples were collected from the antecubital vein at timed intervals after cuff deflation in both methods. It was noted that ischemic -preconditioning prior to prolonged forearm ischemia prevented both endothelial dysfunction and neutrophil activation.

Unfortunately, although pre-conditioning has been extensively studied and has shown to reduce reperfusion injury in both animal and human models, it is difficult to practically apply this in a patient-care setting. This is because the timing of acute cardiac or neurologic ischemic events is difficult to reliably predict. Accordingly, this has generated great interest in a theory known as post-conditioning. Post conditioning or ischemic post-conditioning is a concept whereby short, repetitive ischemic episodes applied during early reperfusion of ischemic myocardium will attenuate reperfusion injury. It appears that both pre-conditioning and post-conditioning target the same pathophysiological mechanism, or share effects on a final common pathway involved in the pathogenesis of reperfusion injury. In a recent study, the effects of ischemic post-conditioning were compared to ischemic preconditioning in the coronary circulation of an animal model. An open chest, left anterior descending coronary artery occlusion model was used in 29 dots (10 controls, 9 preconditioning, and 10 post-conditioning). When compared to controls, both interventions showed protective myocardial effects. The strategy of post-conditioning had comparable results to ischemic preconditioning regarding reduction in infarct size.

Endothelial dysfunction is on of the signs of early atherosclerosis, and also a major component of ischemia-reperfusion injury. Several factors affect endothelial function, but the presence of reactive oxygen species in the vessel wall and the ability of endothelium to generated nitric oxide (NO) seem to be the most important determinants of endothelial function. Due to abnormalities in NOS, the generation of free oxygen radicals increases, and the level of NO decreases during an ischemic episode. This leads to significant alterations in the endothelial function. Under ischemic conditions, nitric oxide synthase produces superoxide (.O2-) in excess of nitric oxide (NO). Superoxide can react with the surrounding nitric oxide to produce a potent oxidizing agent, peroxynitrite (ONOO-). These oxygen radicals are thought to contribute to the development of ischemia-reperfusion injury in humans. NO has been shown to play a significant role in reducing reperfusion injury in humans. The group from our institution demonstrated this where reperfusion injury in the forearm of human subjects was attenuated by the administration of tetrahydrobiopterin (BH4), a cofactor for NOS that leads to the production of NO (unpublished data, Baballiaros et al.). The time course for oxidative marker expression, such as NO, after ischemia-reperfusion injury is expected to occur as early as 2.5 to 5 minutes after reperfusion. Several studies have examined the time course of NO, nitrosyl hemoglobin, glutathione reduction-oxidation, and hydro peroxides. In a study conducted by Mochizuki et al, describing an arterial flow mediated dilation model, NO attained a peak value with a first-order time delay and the peak level NO concentration was linearly correlated with perfusion rate in each vessel. It must be noted, however, that the peak and duration of the levels are somewhat variable and depend on perfusion flow and the diameter of the vessel.

Endothelial function can be non-invasively evaluated using Brachial (or Radial) artery reactivity testing (BART) as a measure of flow-mediated dilation (FMD). Since it's beginnings in 1989, the study of FMD has now taken on an expanded role in the understanding of endothelial physiology. FMD is an endothelial dependent process that reflects relaxation of a conduit artery when exposed to shear stress. Increased flow, and thereby increased shear stress, through the brachial artery occurs after post occlusive reactive hyperemia. Several studies have suggested that the maximal increase in diameter occurs after approximately 60 seconds after the release of the occlusive cuff or after 45-60 seconds after peak reactive hyperemia blood flow. The increase in diameter at this time is prevented by the NO synthase inhibitor, N-G monomethyl-L-arginine, indicating that it is an endothelial dependent process mediated by NO. Other measures of vasodilator response include time to maximum response, duration of the vasodilator response, and the area under the dilation curve .An impairment of endothelial function, via FMD assessment by BART, has been shown to correlate with risk factors for coronary artery disease (smoking, hyperlipidemia, diabetes mellitus) and adverse cardiovascular events.

Currently, there is data that shows the benefit of post-conditioning in reducing reperfusion injury in animal models only. However the use of post-conditioning in humans to reduce reperfusion injury has not been well investigated.Given that endothelial dysfunction is a significant component of reperfusion injury, we propose to examine the effects of post-conditioning on a reperfusion injury by using BART. This study will act as a pilot by which we can compare the results of Post-conditioning to preconditioning to reduce the reperfusion injury with BART in a human reperfusion injury model. The clinical relevance of this study is paramount. If it can be shown that post-conditioning attenuates reperfusion injury in humans, as assessed by BART a larger scale trial to assess post-conditioning on prevention of ischemia reperfusion injury in humans will be necessary. Furthermore, this allows for a possible therapeutic application in the clinical setting, such as potentially providing post-conditioning measures to patients undergoing percutaneous coronary intervention for abruptly occluded coronary arteries. Attenuation of reperfusion injury may further reduce the associated morbidity and mortality of acute coronary ischemic events.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers between the ages of 18 and 35.
* Able to give informed and witnessed consent.
* Don't have the following risk factor

  1. Non smoker
  2. LDL<180, HDL>30, TG<200 or LDL/HDL<6.0
  3. Does not have diabetes mellitus .
  4. BP < 135/85
  5. Do not have family history defined as a parent or sibling with coronary disease diagnosed before age 40. .

Exclusion Criteria:

* Patients with significant medial illness for which they are receiving continued monitoring or treatment, known cardiovascular disease, or risk factors for coronary artery disease are excluded. These risk factors include

  1. Smoking
  2. Hyperlipidemia defined as and LDL>180, HDL<30, TG>200 or LDL/HDL>6.0
  3. Diabetes mellitus
  4. Hypertension,
  5. Strong family history defined as a parent or sibling with coronary disease diagnosed before age 40.

The exclusion criteria are to prevent the confounding effects of atherosclerosis or other medical conditions in our study.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20
Dates: Start 2006-05; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Helmy, MD, Principal Investigator — Emory University; Arshed Ali Quyyumi, MD, Principal Investigator — Emory University; Muhammad Amer, MD, Study Director — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States